CLINICAL TRIAL: NCT01822834
Title: Bronchiectasis and NTM Research Registry
Status: Recruiting | Type: Observational
Sponsor: COPD Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: BRR
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Non-CF Bronchiectasis; Nontuberculosis Mycobacteria (NTM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-CF Bronchiectasis Patients with or without NTM: Patients over the age of 18 with non-CF Bronchiectasis with or without Nontuberculosis Mycobacteria (NTM).
- Nontuberculosis Mycobacteria (NTM): Patients over the age of 18 with Nontuberculosis Mycobacteria (NTM)

SUMMARY:
The Bronchiectasis Research Registry is a consolidated database of non-cystic fibrosis (non-CF) Bronchiectasis and Nontuberculosis Mycobacteria (NTM) patients from multiple clinical institutions.

DETAILED DESCRIPTION:
The Bronchiectasis Research Registry is a consolidated database of non-cystic fibrosis (non-CF) Bronchiectasis and Nontuberculosis Mycobacteria (NTM) patients from multiple clinical institutions. The goal of the Bronchiectasis Research Registry is to support collaborative research and assist in the planning of multi-center clinical trials for the treatment of NTM and non-CF Bronchiectasis, a progressive, non-curable disease of the lungs, which afflicts thousands of patients. The Registry will also be used to provide better insight into the study of the different types of Bronchiectasis, as well as the pathophysiology of the disorder. In 2012, in collaboration with NTM Info and Research, Inc (NTMir) and the consortium members, the COPD Foundation expanded the Bronchiectasis Research Registry to enroll patients with "non tuberculous mycobacteria (NTM) only". Prior to this time, the registry included individuals with Bronchiectasis, with or without NTM.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* non-CF Bronchiectasis
* Nontuberculosis Mycobacteria (NTM)

Exclusion Criteria:

* Under the age of 18
* CF Bronchiectasis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 with non-CF Bronchiectasis and/or Nontuberculosis Mycobacteria (NTM).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-01; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Patient Recruitment and Data analysis | December 2050
  The COPD Foundation expects to assist at least 4 researchers (with patient recruitment and/or data analysis) annually.

CONTACTS AND LOCATIONS:
Locations (1):
- COPD Foundation, Washington D.C., District of Columbia, United States